CLINICAL TRIAL: NCT05031130
Title: The Effects of Empowerment Program Integrated With Family Support on Maternal Self-Esteem and Quality of Life Among Pregnant Adolescents in Palestine: A Randomized Controlled Trial
Brief Title: Effects of Empowerment Program Integrated With Family Support on Maternal Self-esteem and Quality of Life Among Palestinian Pregnant Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Shurouq Ghalib Mousa Qadous, Principle Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PSU IRB 2021-St-Nur 009
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pregnant Adolescents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): For the control group, the researcher will provide routine care to pregnant adolescents.
- Experimental group (Experimental): For the experimental group, the researcher will provide the empowered program integrated with family support plus routine care.
  Interventions: Other: Empowered program integrated with family support

INTERVENTIONS:
Other: Empowered program integrated with family support — The empowered program integrated with family support is an intervention consisted of five steps that will be given when pregnant adolescents on gestational age 32 or 33 weeks the second meeting will be when the pregnant adolescents on gestational age 34 or 35 weeks.
  Arms: Experimental group

SUMMARY:
Adolescent pregnancy leads to increase risks and complications for the adolescent mother and her newborn. This study aims to examine the effects of empowerment program integrated with family support on maternal self-esteem and quality of life among Palestinian pregnant adolescents. A randomized controlled single-blind trial, pretest-posttest controlled group design will be conducted with 62 participants ( control group =31, experimental group = 31). Research instruments will include the instruments for data collection, instruments for research intervention, and control instruments for intervention evaluation. The instruments for data collection will be consists of a demographic data form, Maternal Self-Report Inventory (MSRI), and WHO quality of life-BREF (WHOQoL-BREF, 1997). The empowerment program integrated with family support will be the research intervention instruments and included five steps; step 1: building relationships and creating collaboration, step 2: discovering reality, step 3: critical reflection, step 4: taking charge, and step 5: holding on. Control instruments through Family Support Questionnaire (FSQ) will be used to evaluate the effectiveness of the intervention program. Data will be analyzed using mean and standard deviations, frequency distribution, percentage, and chi-square test, and t-test. This program is expected to guide nurses to empower pregnant adolescents in enhancing maternal self-esteem and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 15 to 20 years.
2. First-time pregnant.
3. Have a single fetus.
4. Gestational age 32 or 33 weeks.
5. Medical history free from diseases such as diabetes mellitus (DM), hypertension, urinary tract infections (UTIs), heart disease, and thyroid disease.
6. Free of complications during the present pregnancy such as preterm labor and gestational hypertension.
7. Have more than check answers on the perinatal screening depression checklist (adopted from Edinburgh Postnatal Depression Scale).
8. Having their own family member (pregnant adolescents' husband, own mother, mother-in-law, her sister, or sister-in-law) during giving the intervention.
9. Able to read, write, and communicate clearly in the Arabic language.
10. Living in Nablus City.

The family member will be included in any of the following criteria are present.

1. Being with the pregnant adolescent during the intervention and continue giving support at home.
2. The available phone number for contact while family members are at home.

Exclusion Criteria:

1. Pregnant adolescents who experience any serious obstetric complications during the study such as preterm labor, gestational hypertension, and bleeding disorders.
2. Pregnant adolescent who is not able to follow or complete the intervention program.
3. Family member who is unable to accompany the pregnant adolescent during the intervention delivery at the primary health care clinic.
4. Family member who is unable to give social support to the pregnant adolescent at home.
5. Pregnant adolescents or family members in case one of them withdraws from the study the other will be excluded from the study.

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Maternal Self-Esteem (MSE) | Measure MSE at 32 weeks gestation or 33 weeks gestation (Preintervention)
  Used Maternal Self Report Inventory-Short Form (MSRI-SF)
Quality of Life (QoL) | Measure QoL at 32 weeks gestation or 33 weeks gestation (Preintervention)
  Used World Health Organization Quality of Life- BREF (WHOQoL-BREF)
Maternal Self-Esteem (MSE) | Measure MSE at 36 weeks gestation or 37 weeks gestation (Postintervention)
  Used Maternal Self Report Inventory-Short Form (MSRI-SF)
Quality of Life (QoL) | Measure QoL at 36 weeks gestation or 37 weeks gestation (Postintervention)
  Used World Health Organization Quality of Life- BREF (WHOQoL-BREF)

CONTACTS AND LOCATIONS:
Overall Officials: Shurouq Qadous, Principal Investigator — Prince Songkla University
Locations (1):
- Shurouq Ghalib Qadous, Nablus, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qadous SG, Chunuan S, Chatchawet W. Effectiveness of a nurse-led family empowerment program to improve the quality of life among pregnant adolescents: A randomized controlled trial. Int J Gynaecol Obstet. 2025 Feb;168(2):716-723. doi: 10.1002/ijgo.15881. Epub 2024 Sep 3. PMID 39224986